CLINICAL TRIAL: NCT01081054
Title: Randomized Trial Comparing Two Treatment Strategies for Acute Diverticulitis. Hospitalization or Ambulatory Antibiotic Treatment
Brief Title: Hospitalization or Ambulatory Treatment of Acute Diverticulitis
Acronym: 01DIVER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Universitari de Bellvitge (Other)
Responsible Party: Principal Investigator, Sebastiano Biondo, S. Biondo, MD, PhD, Colorectal Unit, Department of Surgery, Hospital Universitari de Bellvitge
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01DIVER; 2008-008452-17 (EudraCT Number)
Record Dates: First submitted 2010-03-04; First posted 2010-03-05 (Estimated); Last update posted 2012-06-12 (Estimated); Status verified 2012-06

CONDITIONS: Diverticulitis
Keywords: Diverticulitis; Not complicated diverticulitis
MeSH Terms: conditions — Diverticulitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ambulatory Treatment (Other): Patients are treated ambulatory with oral antibiotic for 10 days; for the first five days these patients are contacted by telephone daily to progress oral intake.
  Interventions: Other: Ambulatory versus hospitalisation
- Hospital treatment (Active Comparator): Patients are hospitalized and treated with antibiotic, for the first days by endovenous antibiotic and with diet progression orally.
  Interventions: Other: Ambulatory versus hospitalisation

INTERVENTIONS:
Other: Ambulatory versus hospitalisation — Patients are treated with the same antibiotic agent, the difference between the two arms is endovenous treatment for hospitalized patients for the first days till oral feeding. The ambulatory group starts directly with orally administered antibiotic treatment.

SUMMARY:
The purpose of 01DIVER is to evaluate efficacy and safety of a home treatment protocol for non complicated diverticulitis compared with management in the hospital. The hypothesis is that a ambulatory treatment with oral antibiotic and progressive introduction of diet is not inferior to the conservative management in hospital in patients with acute not complicated sigmoid diverticulitis, shown by contrast enhanced CT scan. Patients are prospectively randomized to conservative antibiotic treatment either to ambulatory or to hospital treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age older than 18 years
* Diagnosis of mild diverticulitis by abdominal computerized tomography
* Signed informed consent

Exclusion Criteria:

* Severe diverticulitis
* Informed consent not signed
* Suspicion of colon cancer
* Pneumoperitoneum
* Intolerance for oral feeding
* Antibiotics for diverticulitis in the last month
* Immunosuppression
* Pregnancy or lactation
* Severe (decompensated) other illness
* Psychological or social problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2009-09; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Treatment failure | 30 days
  Failure of the conservative treatment within 30 days after randomization which consists in one or more of the mentioned signs: persistent or increasing pain, treatment resistant fever, intestinal oclusion, necesity to drain a new intra-abdominal abscess, indication for surgery, mortality.

SECONDARY OUTCOMES:
Recurrence, quality of life, costs | 30 days
  Recurrence of diverticulitis within 30 days; quality of life and patient satisfaction is asessed comparing management with and without admittance to the hospital and costs are calculated for the treatment in both regimens.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastiano Biondo, MD, PhD, Principal Investigator — Hospital Universitari de Bellvitge
Locations (5):
- Spain (5):
  - Hospital Universitari de la Vall d´Hebron, Barcelona, Barcelona
  - Hospital Universitari Bellvitge, Colorectal Unit, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitari de Girona Doctor Josep Trueta, Girona, Girona
  - Hospital Virgen del Camino, Pamplona, Navarre
  - Hospital Clinico Universitario De Valencia, Valencia, Valencia